CLINICAL TRIAL: NCT06804629
Title: Acute and Chronic Effects of Guidelines-Based Resistance Exercise Training Compared to a Low Intensity SHAM Attention Control Among Young Adult Women With Analogue Generalized Anxiety Disorder: A Protocol for a Randomized Controlled Trial.
Brief Title: The Resistance Exercise Training for Worry Trial: Replication and Expansion
Acronym: RETRAIN REP-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Taighde Éireann - Research Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017_03_18_EHS_new; GOIPG/2023/4158 (Other Grant/Funding Number: Taighde Éireann - Research Ireland)
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Analogue Generalized Anxiety Disorder
Keywords: Analogue Generalized Anxiety Disorder; Young adults; Female; Worry; Strength training; Resistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial of ten weeks of moderate-to-high compared to low intensity SHAM resistance exercise training among young adult women with analogue Generalized Anxiety Disorder
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator was blinded to group allocation and performed blinded outcome analyses. Blinding of the investigators who supervised the resistance exercise training sessions was not possible. Participants were not informed of whether they were randomized to an intervention or control group, or of the study hypothesis. At baseline, each participant received an identification number which remained the same throughout the trial. Information that could potentially identify any participant was removed from the working dataset after full data extraction from Qualtrics, such that participants could not be identified based on personal characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate-to-High Intensity Resistance Exercise Training (Experimental): Moderate-to-high intensity, guidelines-based resistance exercise training completed at 70-80% of the estimated one-repetition maximum
  Interventions: Behavioral: Moderate-to-High Intensity Resistance Exercise Training
- Low Intensity SHAM Resistance Exercise Training Attention Control (Sham Comparator): Low intensity SHAM Resistance Exercise Training completed at 20% of the estimated one-repetition maximum
  Interventions: Behavioral: Low Intensity SHAM Resistance Exercise Training Attention Control

INTERVENTIONS:
Behavioral: Moderate-to-High Intensity Resistance Exercise Training — Resistance exercise training was designed in accordance with World Health Organization and American College of Sports Medicine guidelines. The eight-week, twice-weekly intervention was designed such that moderate-to-high intensity participants could achieve two sets of 8-12 repetitions of the eight exercises before volitional fatigue, a deterioration in lifting form, or failure to complete a repetition, using loads of approximately 70-80% of their estimated one-repetition maximum. Completed in the following order, the exercises were: barbell back squat, barbell bench press, hexagon bar deadlift, barbell bent over row, dumbbell lunges, seated dumbbell lateral raises, weighted or unweighted abdominal crunches, and seated dumbbell bicep curls. There was one minute of rest between each set, and two minutes of rest between each exercise. If participants could complete two sets of 12 repetitions, load was increased gradually by approximately 5% in the following session.
  Other Names: Strength training; Weight-lifting
  Arms: Moderate-to-High Intensity Resistance Exercise Training
Behavioral: Low Intensity SHAM Resistance Exercise Training Attention Control — The low intensity SHAM condition was matched all features of engagement with the moderate-to-high intensity intervention apart from load, and load progression. Low intensity SHAM participants completed the same program with loads of approximately 20% of their estimated one-repetition maximum. To maintain low intensity, repetitions completed on the main, heavier lifts (i.e., back squat, bench press, deadlift, bent over row) were increased from 10 in one session to 12 in the next; load was then increased by approximately 10% in the following session, and 10 reps were performed again. On the remaining lighter, assistance lifts, eight repetitions were performed per set, then one repetition was added to both sets in each session, and load was increased by the smallest increment possible when two sets of 12 repetitions were performed. Borg's 6-20 rating of perceived exertion scores were used to monitor intensity, such that if scores exceeded 11, load and reps were not progressed.
  Arms: Low Intensity SHAM Resistance Exercise Training Attention Control

SUMMARY:
This protocol details the full methods of a ten-week moderate-to-high intensity, guidelines-based resistance exercise training intervention compared to a low intensity sham attention control among young adult women with analogue Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
A recent clinical trial supported the anxiolytic effects of regularly-performed resistance exercise training compared to a waitlist control among young adults with and without at least subclinical, or analogue, Generalized Anxiety Disorder. Although the evidence to date is promising, waitlist control conditions cannot control for potential social and psychological benefits of engaging with most interventions, including social contact, expectations for improvement, and mastery experiences, which could potentially be achieved from easier activities. Therefore, this trial aims to replicate the previously investigated World Health Organization and American College of Sports Medicine guidelines-based resistance exercise training program, and expand on this research by more rigorously examining the effects on anxiety and worry symptoms, independent of potential social and psychological benefits of engagement with the intervention. Consequently, this trial quantifies the acute and chronic effects of moderate-to-high intensity, guidelines-based resistance exercise training compared to a low intensity SHAM attention control on signs and symptoms of Generalized Anxiety Disorder among at-risk young adult women with Analogue Generalized Anxiety Disorder. This trial consists of a two-week familiarization protocol, eight weeks of formal resistance exercise training, and a one-month post-intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-40y
* Met criteria for analogue Generalized Anxiety Disorder

Exclusion Criteria:

* Medical contraindications to doing resistance exercise training
* Currently involved in formal resistance exercise training
* Currently pregnant or post-partum

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Analogue Generalized Anxiety Disorder Status | Baseline
  Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001)
Analogue Generalized Anxiety Disorder Status | Week 1
  Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001)
Analogue Generalized Anxiety Disorder Status | Week 4
  Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001)
Analogue Generalized Anxiety Disorder Status | Week 8
  Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001)
Analogue Generalized Anxiety Disorder Status | Week 12
  Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001)
Analogue Generalized Anxiety Disorder Status | Baseline
  Penn State Worry Questionnaire of 45 or greater (Meyer et al., 1990)
Analogue Generalized Anxiety Disorder Status | Week 1
  Penn State Worry Questionnaire of 45 or greater (Meyer et al., 1990)
Analogue Generalized Anxiety Disorder Status | Week 4
  Penn State Worry Questionnaire of 45 or greater (Meyer et al., 1990)
Analogue Generalized Anxiety Disorder Status | Week 8
  Penn State Worry Questionnaire of 45 or greater (Meyer et al., 1990)
Analogue Generalized Anxiety Disorder Status | Week 12
  Penn State Worry Questionnaire of 45 or greater (Meyer et al., 1990)
Worry Symptoms | Baseline
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Pre-week 1
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 1
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 2
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 3
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 4
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 5
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 6
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 7
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 8
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)
Worry Symptoms | Week 12
  16-item Penn State Worry Questionnaire (Meyer et al., 1990)

SECONDARY OUTCOMES:
Anxiety Symptoms | Baseline
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Pre-week 1
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 1
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 2
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 3
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 4
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 5
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 6
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 7
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 8
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Week 12
  Trait anxiety was measured using the Trait (STAI-Y2) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Baseline
  State anxiety was measured using the State (STAI-Y1) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Pre-acute resistance exercise bout week 1
  State anxiety was measured using the State (STAI-Y1) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Post-acute resistance exercise bout week 1
  State anxiety was measured using the State (STAI-Y1) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Pre-acute resistance exercise bout week 8
  State anxiety was measured using the State (STAI-Y1) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Anxiety Symptoms | Post-acute resistance exercise bout week 8
  State anxiety was measured using the State (STAI-Y1) subscale of the State-Trait Anxiety Inventory (Spielberger, 2010)
Depressive Symptoms | Baseline
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Pre-week 1
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 1
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 2
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 3
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 4
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 5
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 6
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 7
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 8
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Depressive Symptoms | Week 12
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003)
Mood | Baseline
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Pre-week 1
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 1
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 2
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 3
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 4
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 5
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 6
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 7
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 8
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 12
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Pre-acute resistance exercise bout week 1
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Post-acute resistance exercise bout week 1
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Pre-acute resistance exercise bout week 8
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Post-acute resistance exercise bout week 8
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Analogue Major Depressive Disorder Status | Baseline
  Psychiatric Diagnostic Screening Questionnaire Major Depressive Disorder subscale score of 9 or greater (Zimmerman & Mattia, 2001)
Analogue Major Depressive Disorder Status | Week 1
  Psychiatric Diagnostic Screening Questionnaire Major Depressive Disorder subscale score of 9 or greater (Zimmerman & Mattia, 2001)
Analogue Major Depressive Disorder Status | Week 4
  Psychiatric Diagnostic Screening Questionnaire Major Depressive Disorder subscale score of 9 or greater (Zimmerman & Mattia, 2001)
Analogue Major Depressive Disorder Status | Week 8
  Psychiatric Diagnostic Screening Questionnaire Major Depressive Disorder subscale score of 9 or greater (Zimmerman & Mattia, 2001)
Analogue Major Depressive Disorder Status | Week 12
  Psychiatric Diagnostic Screening Questionnaire Major Depressive Disorder subscale score of 9 or greater (Zimmerman & Mattia, 2001)
Analogue Panic Disorder Status | Baseline
  Psychiatric Diagnostic Screening Questionnaire Panic Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Panic Disorder Status | Week 1
  Psychiatric Diagnostic Screening Questionnaire Panic Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Panic Disorder Status | Week 4
  Psychiatric Diagnostic Screening Questionnaire Panic Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Panic Disorder Status | Week 8
  Psychiatric Diagnostic Screening Questionnaire Panic Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Panic Disorder Status | Week 12
  Psychiatric Diagnostic Screening Questionnaire Panic Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Social Anxiety Disorder Status | Baseline
  Psychiatric Diagnostic Screening Questionnaire Social Anxiety Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Social Anxiety Disorder Status | Week 1
  Psychiatric Diagnostic Screening Questionnaire Social Anxiety Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Social Anxiety Disorder Status | Week 4
  Psychiatric Diagnostic Screening Questionnaire Social Anxiety Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Social Anxiety Disorder Status | Week 8
  Psychiatric Diagnostic Screening Questionnaire Social Anxiety Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Analogue Social Anxiety Disorder Status | Week 12
  Psychiatric Diagnostic Screening Questionnaire Social Anxiety Disorder subscale score of 4 or greater (Zimmerman & Mattia, 2001)
Sleep Quality | Baseline
  Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Sleep Quality | Week 1
  Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Sleep Quality | Week 4
  Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Sleep Quality | Week 8
  Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Sleep Quality | Week 12
  Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Irritability Symptoms | Baseline
  21-item Irritability Questionnaire (Craig et al., 2008)
Irritability Symptoms | Week 1
  21-item Irritability Questionnaire (Craig et al., 2008)
Irritability Symptoms | Week 4
  21-item Irritability Questionnaire (Craig et al., 2008)
Irritability Symptoms | Week 8
  21-item Irritability Questionnaire (Craig et al., 2008)
Irritability Symptoms | Week 12
  21-item Irritability Questionnaire (Craig et al., 2008)
Rumination | Baseline
  Rumination-Reflection Questionnaire (Trapnell and Campbell, 1999)
Rumination | Week 1
  Rumination-Reflection Questionnaire (Trapnell and Campbell, 1999)
Rumination | Week 4
  Rumination-Reflection Questionnaire (Trapnell and Campbell, 1999)
Rumination | Week 8
  Rumination-Reflection Questionnaire (Trapnell and Campbell, 1999)
Rumination | Week 12
  Rumination-Reflection Questionnaire (Trapnell and Campbell, 1999)
Cognitive Functioning | Baseline
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Pre-acute resistance exercise bout week 1
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Post-acute resistance exercise bout week 1
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Pre-acute resistance exercise bout week 8
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Post-acute resistance exercise bout week 8
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Week 8
  Stroop Colour and Word Test (Williams et al., 1996)
Cognitive Functioning | Baseline
  Trail Making Test (Tombaugh, 2004)
Cognitive Functioning | Pre-acute resistance exercise bout week 1
  Trail Making Test (Tombaugh, 2004)
Cognitive Functioning | Post-acute resistance exercise bout week 1
  Trail Making Test (Tombaugh, 2004)
Cognitive Functioning | Pre-acute resistance exercise bout week 8
  Trail Making Test (Tombaugh, 2004)
Cognitive Functioning | Post-acute resistance exercise bout week 8
  Trail Making Test (Tombaugh, 2004)
Cognitive Functioning | Week 8
  Trail Making Test (Tombaugh, 2004)
Resistance Exercise Expectations | Baseline
  15-item Expected Psychological Outcomes of Resistance Exercise Training (EPO-RET) questionnaire, derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants were asked "For each of the below outcomes, think about how you would expect to feel after completing a resistance exercise program (2 sessions per week for 8-12 weeks) relative to how you typically feel".
Resistance Exercise Expectations | Week 1
  15-item Expected Psychological Outcomes of Resistance Exercise Training (EPO-RET) questionnaire, derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants were asked "For each of the below outcomes, think about how you would expect to feel after completing a resistance exercise program (2 sessions per week for 8-12 weeks) relative to how you typically feel".
Resistance Exercise Expectations | Week 4
  15-item Expected Psychological Outcomes of Resistance Exercise Training (EPO-RET) questionnaire, derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants were asked "For each of the below outcomes, think about how you would expect to feel after completing a resistance exercise program (2 sessions per week for 8-12 weeks) relative to how you typically feel".
Resistance Exercise Expectations | Week 8
  15-item Expected Psychological Outcomes of Resistance Exercise Training (EPO-RET) questionnaire, derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants were asked "For each of the below outcomes, think about how you would expect to feel after completing a resistance exercise program (2 sessions per week for 8-12 weeks) relative to how you typically feel".
Resistance Exercise Expectations | Week 12
  15-item Expected Psychological Outcomes of Resistance Exercise Training (EPO-RET) questionnaire, derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants were asked "For each of the below outcomes, think about how you would expect to feel after completing a resistance exercise program (2 sessions per week for 8-12 weeks) relative to how you typically feel".
Resistance Exercise Expectations | Pre-acute resistance exercise bout week 1
  15-item Expected Psychological Outcomes of Acute Resistance Exercise (EPO-ARE) derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants are asked to "think about how you would expect to feel after one resistance exercise workout relative to how you typically feel".
Resistance Exercise Expectations | Post-acute resistance exercise bout week 1
  15-item Expected Psychological Outcomes of Acute Resistance Exercise (EPO-ARE) derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants are asked to "think about how you would expect to feel after one resistance exercise workout relative to how you typically feel".
Resistance Exercise Expectations | Pre-acute resistance exercise bout week 8
  15-item Expected Psychological Outcomes of Acute Resistance Exercise (EPO-ARE) derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants are asked to "think about how you would expect to feel after one resistance exercise workout relative to how you typically feel".
Resistance Exercise Expectations | Post-acute resistance exercise bout week 8
  15-item Expected Psychological Outcomes of Acute Resistance Exercise (EPO-ARE) derived from the Expected Psychological Outcomes of Exercise Questionnaire (Lindheimer et al., 2020). Participants are asked to "think about how you would expect to feel after one resistance exercise workout relative to how you typically feel".
Physical Activity | Baseline
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Pre-week 1
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 1
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 2
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 3
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 4
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 5
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 6
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 7
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 8
  7-day Physical Activity Recall (Blair et al., 1985)
Physical Activity | Week 12
  7-day Physical Activity Recall (Blair et al., 1985)
Muscle-Strengthening Exercise Activity | Baseline
  Muscle-Strengthening Exercise Questionnaire - Short Version (Shakespear-Druery et al., 2022)
Muscle-Strengthening Exercise Activity | Week 1
  Muscle-Strengthening Exercise Questionnaire - Short Version (Shakespear-Druery et al., 2022)
Muscle-Strengthening Exercise Activity | Week 4
  Muscle-Strengthening Exercise Questionnaire - Short Version (Shakespear-Druery et al., 2022)
Muscle-Strengthening Exercise Activity | Week 8
  Muscle-Strengthening Exercise Questionnaire - Short Version (Shakespear-Druery et al., 2022)
Muscle-Strengthening Exercise Activity | Week 12
  Muscle-Strengthening Exercise Questionnaire - Short Version (Shakespear-Druery et al., 2022)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Herring, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Primary outcome data will be made available for five years at six months following publication of primary outcome summary data. Secondary outcome data will be made available for five years at six months following publications of secondary outcome summary data.
Access Criteria: Proposals should be directed to matthew.herring@ul.ie. To gain access, data requestors will need to sign a data access agreement.